CLINICAL TRIAL: NCT05518227
Title: Patient Satisfaction and Visual Outcomes After Bilateral PanOptix Implantation in Patients With Previous Multifocal Contact Lens
Status: Terminated | Type: Observational
Why Stopped: recruitment slow
Sponsor: Vivid Laser Center (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: RB-22-001
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- The Clareon™ PanOptix™ Trifocal (toric and non-toric models): Bilateral implantation with the Clareon PanOptix Trifocal (toric and non-toric models)
  Interventions: Device: The Clareon™ PanOptix™ Trifocal (toric and non-toric models)

INTERVENTIONS:
Device: The Clareon™ PanOptix™ Trifocal (toric and non-toric models) — Bilateral implantation with the Clareon PanOptix Trifocal (toric and non-toric models)

SUMMARY:
To evaluate spectacle independence and patient satisfaction and visual outcomes after bilateral PanOptix implantation in patients with previous multifocal contact lens experience.

DETAILED DESCRIPTION:
This study is a single-arm unmasked clinical evaluation study of patient satisfaction after successful bilateral cataract surgery. Subjects will be assessed pre-operatively, operatively and at 1 day, 1 week and 3 months post-operatively. Clinical evaluations will include administration of a visual disturbance questionnaire (QUVID), and a satisfaction questionnaire (IOLSAT), as well as measurement of bilateral visual acuity and manifest refraction.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Adult cataract patients undergoing uncomplicated cataract surgery with Clareon PanOptix IOL implantation (non-toric/toric).
* Visually significant cataracts bilaterally.
* History of successful soft multifocal contact lens use in the past (within ≤ last 5 years).
* Healthy ocular exam.
* Gender: Males and Females.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Previous monovision patients.
* Ocular comorbidity that might hamper post operative visual acuity (Uveitis, Keratoconus, Retinopathies, Glaucoma).
* Previous ocular or refractive surgery.
* Expected monocular post-op distance VA worse than 20/25 (Snellen) in either eye.
* Refractive lens exchange.
* Angle kappa measurement in a single eye over 0.6 mm.
* Irregular corneal astigmatism or ectasia.
* Difficulties comprehending written or spoken English language.
* Patients with physical or intellectual disability (e.g. Down's Syndrome, Parkinson's Disease; unable to fixate).
* Severe/uncontrolled Ocular surface disease/Dry Eye Disease.
* Intraoperative complications during procedure.
* Visual expectations exceed outcomes.
* Strabismus (with or without amblyopia).

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants will be presenting for cataract surgery who are interested in a reduced dependence on spectacles for near, intermediate, and distance vision, and who are considered appropriate candidates for trifocal lens implantation.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Satisfaction questionnaire | 3 months postoperative
  The Intraocular Lens Satisfaction questionnaire (IOLSAT). Lower scores indicate higher spectacle independence and satisfaction.

SECONDARY OUTCOMES:
Binocular uncorrected distance visual acuity (6m) | 3 months postoperative
Binocular uncorrected intermediate visual acuity (60 cm) | 3 months postoperative
Binocular uncorrected near visual acuity (40 cm) | 3 months postoperative
Binocular corrected distance visual acuity (6m) | 3 months postoperative
Binocular distance corrected intermediate visual acuity (60 cm) | 3 months postoperative
Binocular distance corrected intermediate visual acuity (40 cm) | 3 months postoperative
Manifest refraction | 3 months postoperative
Spectacle independence | 3 months postoperative
  The Intraocular Lens Satisfaction questionnaire (IOLSAT). Lower scores indicate higher spectacle independence and satisfaction.

OTHER OUTCOMES:
Binocular distance corrected intermediate visual acuity (33 cm) | 3 months postoperative
Visual disturbances questionnaire | 3 months postoperative
  Questionnaire for Visual Disturbances (QUVID). Lower scores indicate less frequent, severe, or bothersome visual disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Baldassare, MD, Principal Investigator — Vivid Laser Center
Locations (1):
- Vivid Laser Center, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No